CLINICAL TRIAL: NCT06361238
Title: Perioperative Application of Liraglutide for the Prevention of Postoperative Delirium Among Elderly Patients with Type 2 Diabetes Undergoing Cardiac Surgery: a Single-Center Randomized Controlled Study
Brief Title: Liraglutide in Preventing Delirium in Diabetic Elderly After Cardiac Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-LCYJ-PY-21
Record Dates: First submitted 2024-03-19; First posted 2024-04-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Delirium, Postoperative
MeSH Terms: conditions — Emergence Delirium | interventions — Liraglutide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liraglutide Group (Experimental): Subcutaneous injection of liraglutide
  Interventions: Drug: Liraglutide injection
- Vehicle Group (Placebo Comparator): Subcutaneous injection of vehicle
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: Liraglutide injection — Subcutaneous injection of liraglutide: 0.6 mg administered the day before surgery, 1.8 mg administered post-anesthesia induction on the day of surgery, followed by 0.6 mg daily for the first three postoperative days.
  Other Names: Victoza
  Arms: Liraglutide Group
Drug: Placebo injection — Subcutaneous injection of Placebo: the same volume as liraglutide administrated at the corresponding times.
  Other Names: Normal saline
  Arms: Vehicle Group

SUMMARY:
This study aims to clarify the preventive effect of perioperative liraglutide application on postoperative delirium in elderly patients with Type 2 diabetes undergoing cardiac surgery.

DETAILED DESCRIPTION:
Delirium is the most prevalent neurological complication following cardiac surgery. It is characterized by an acute and fluctuating disturbance in consciousness, attention, and cognitive function. The incidence of delirium post-cardiac surgery ranges between 11% and 46%. It is closely linked to increased postoperative mortality, extended hospital stays, higher healthcare costs, and long-term cognitive impairment. Currently, it is widely recognized that the development of delirium is influenced by multiple factors, including advanced age, diabetes, surgical and anesthetic techniques, depression, baseline cognitive function, and infections, among others.

Inflammatory responses, crucial for protecting against external or internal threats, can, following surgery, lead to neuroinflammation and neurological damage due to elevated postoperative inflammatory markers and blood-brain barrier disruption. The involvement of microglia and astrocytes, key players in the central nervous system's immune response, has been identified in mediating postoperative delirium, making them potential targets for prevention.

Liraglutide, a Glucagon-like peptide-1 receptor agonist primarily used for treating Type 2 diabetes, has shown promise in mitigating neurocognitive damage associated with diabetes and Alzheimer's disease, suggesting its potential in preventing postoperative delirium in cardiac surgery patients with Type 2 diabetes. Preliminary animal studies and a randomized controlled trial indicate that perioperative liraglutide application could reduce the incidence of postoperative delirium by inhibiting glial activation and the subsequent neuroinflammatory response. However, differences in patient demographics, disease severity, and dosing in previous studies highlight the need for further investigation.

The study aims to investigate whether the perioperative administration of liraglutide can prevent the onset of postoperative delirium in elderly patients with Type 2 diabetes undergoing cardiac surgery. Secondary objectives include assessing the impact on the severity and duration of delirium, cognitive function, anxiety, depression, cardiac function, cardiovascular events, ICU stay, mechanical ventilation duration, and levels of serum markers for brain injury, inflammation, myocardial damage, and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years
2. Type 2 diabetes
3. Patients undergoing elective cardiac surgery

Exclusion Criteria:

1. History of neurological or psychiatric disorders, such as schizophrenia, epilepsy, Parkinson's disease, severe dementia, etc
2. Patients with communication difficulties, such as severe visual, auditory, or speech impairments
3. History of central nervous system damage or surgery
4. Cardiac function NYHA Class IV
5. Severe liver dysfunction (Child-Pugh Class C)
6. Severe renal failure requiring renal replacement therapy
7. History of pancreatitis
8. Type 1 diabetes
9. Patients whose blood sugar is difficult to control within 4-8 mmol/L during the screening period
10. Patients with medullary thyroid carcinoma or a family history of it
11. Pregnant or breastfeeding women
12. Intolerance or allergy to liraglutide
13. Previous use of GLP-1A and SGLT2i
14. Patients who refuse to sign the informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of delirium | One day before surgery and within the first seven days after surgery.
  Confusion Assessment Method (CAM), or its variant for the Intensive Care Unit, known as CAM-ICU, is the tool used to assess the incidence of delirium. For CAM, the scale ranges from a minimum value of 11 to a maximum of 44, with higher scores indicating a worse outcome. In contrast, CAM-ICU does not utilize a numerical scale; it is a qualitative assessment designed to evaluate confusion without assigning specific values.

SECONDARY OUTCOMES:
The severity of delirium | One day before surgery and within the first seven days after surgery.
  The CAM-Severity Scale (CAM-S), available in both short-form and long-form versions, serves as a tool for assessing the severity of delirium. The scale extends from 0 to 7 in its short-form and from 0 to 19 in its long-form. Higher scores on the CAM-S are indicative of more severe outcomes.
Cognitive function | One day before surgery; one week after surgery or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  Minimum Mental State Examination (MMSE) is the tool used to assess cognitive function. The scale extends from 0 to 30, with higher scores indicating a better outcome.
Anxiety | One day before surgery; one week after surgery or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  Generalized anxiety disorder-7 (GAD-7) is the tool used to assess anxiety. The scale extends from 0 to 21, with higher scores indicating a worse outcome.
Depression | One day before surgery; one week after surgery or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  Patient Health Questionnaire-9 (PHQ-9) is the tool used to assess depression. The scale extends from 0 to 27, with higher scores indicating a worse outcome.
Duration of ICU stay | The time from transfer into the ICU to discharge from the ICU, assessed up to 12months.
  By retrieving the Hospital Information System and ICU special care sheet
Mechanical ventilation time | The time from tracheal intubation to the removal of the tracheal tube, assessed up to 12months.
  By retrieving the Hospital Information System and ICU special care sheet
Duration of hospital stay | The time from hospital admission to discharge, assessed up to 12months.
  By retrieving the Hospital Information System
In-hospital mortality | The time from hospital admission to discharge, assessed up to 12months.
  By retrieving the Hospital Information System
Incidence of adverse events | One day preoperatively to three days Postoperatively.
  By retrieving the Hospital Information System, ICU special care sheet and follow-up
Rate of major cardiovascular adverse events | Within 1 year post-surgery (including cardiovascular death, myocardial infarction, and stroke)
  By retrieving the Hospital Information System, ICU special care sheet and follow-up
Serum levels of NSE | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of CRP | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of IL-1α | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of TNF-α | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of C3 | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of LDH | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of CK | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of CK-MB | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of AST | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of cTNT | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of BNP | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of C1q | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of IL-1β | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of IL-6 | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Serum levels of S100β | One day preoperatively; immediately after admission to ICU; 3 days and 7 days postoperatively
  ELISA
Left Ventricular Posterior Wall Thickness in Diastole (LVPWTd) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the LVPWTd.
Left Ventricular End-Diastolic Dimension (LVDd) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the LVDd.
Left Ventricular End-Systolic Diameter (LVDs) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the LVDs.
Left Atrial Diameter (LAD) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the LAD.
Ejection Fraction (EF) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the EF.
Fractional Shortening (FS) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the FS.
Early Diastolic Velocity/Atrial Diastolic Velocity (E/A) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the E/A.
Interventricular Septum Thickness in Diastolic (IVSTd) | One day preoperatively; One week postoperatively or at the date of discharge; and at 3 months, 6 months, and 1 year postoperatively.
  The echocardiography is used to assess the IVSTd.

CONTACTS AND LOCATIONS:
Overall Officials: Dongjin Wang, PhD，MD, Principal Investigator — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Wenxue liu, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No